CLINICAL TRIAL: NCT07402889
Title: Adaptation and Validity of the Lithuanian Version of the Baecke Physical Activity Questionnaire
Status: Enrolling by invitation | Type: Observational
Sponsor: Ernesta Aukštuolytė (Other)
Responsible Party: Sponsor-Investigator, Ernesta Aukštuolytė, PhD student, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Other Study IDs: BE-2-143
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Questionnaires; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group - Questionnaire Completion
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No interventions

SUMMARY:
The aim of this study is to adapt the Baecke Questionnaire of Habitual Physical Activity for use in Lithuania.

Individuals who meet the following criteria may participate in this study:

Adults aged 18 years or older. Native Lithuanian speakers. Willingness to participate in the study by signing an informed consent form.

If you agree to take part in this study, you will be asked to visit the Department of Sports Medicine of the Lithuanian University of Health Sciences (Eivenių st. 2, Kaunas) twice. During the first visit, you will be asked to complete the Baecke Questionnaire of Habitual Physical Activity and the International Physical Activity Questionnaire. During height and weight measurements, you will be asked to remove your shoes and outer clothing. After one week, you will be asked to return for a follow-up visit, during which you will complete the Baecke Questionnaire of Habitual Physical Activity again.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older. Native Lithuanian speakers. Willingness to participate in the study by signing an informed consent form.

Exclusion Criteria:

none

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants will include women and men aged ≥18 years.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2029-02-02 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
Baecke Questionnaire of Habitual Physical Activity - test-retest reliability | 1 week between baseline and follow-up administration
  The primary outcome is the consistency of responses to the Baecke Questionnaire of Habitual Physical Activity when completed by the same participants one week apart, to assess the reliability of the adapted Lithuanian version.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant privacy and confidentiality.

REFERENCES:
- [Background] Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. Am J Clin Nutr. 1982;36(5):936-942. doi:10.1093/ajcn/36.5.936